CLINICAL TRIAL: NCT01241006
Title: A Randomized Double-Blind Controlled Trial of Single Oral Dose Dexamethasone Versus Five Days of Oral Prednisone in Acute Mild to Moderate Adult Asthma
Brief Title: Single Oral Dose of Dexamethasone Versus Five Days of Prednisone in Adult Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alameda County Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Rehrer, Chairman of ACMC Emergency Department, Alameda County Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB10-08103G
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Reactive Airway Disease
Keywords: Relapse; Corticosteroids
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Recurrence | interventions — Dexamethasone; Calcium Dobesilate; Prednisone; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Single dose of Dexamethasone 12 mg PO and 4 days of placebo capsules
  Interventions: Drug: Dexamethasone
- Prednisone (Active Comparator): Prednisone 60mg PO capsules for 5 days
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 12mg PO single dose x 1 Placebo 1 capsule PO for 4 days
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Prednisone — Prednisone 60mg PO q day for 5 days
  Other Names: Glucocorticoid
  Arms: Prednisone

SUMMARY:
This study seeks to compare the effectiveness of a single dose of oral dexamethasone versus 5 days of oral prednisone in the treatment of mild to moderate asthma exacerbations to prevent relapse with an unscheduled return visit to a health care provider for additional asthma treatment within 14 days. The investigators hypothesize that the two treatments will be equally effective in relapse prevention.

DETAILED DESCRIPTION:
Dexamethasone and Prednisone are both systemic corticosteroids. The study will compare a single dose of oral dexamethasone to 5 days of oral prednisone in the treatment of asthma. Oral corticosteroids are commonly prescribed following an asthma exacerbation as it has been demonstrated that these medications prevent relapse.

Oral prednisone is the most common corticosteroid prescribed for asthma relapse prevention. The half life is around 4 hours and is typically prescribed for minimally 5 days.

The study is evaluating the efficacy of a single dose of dexmethasone. The drug's efficicacy has been shown to be longer acting and up to 72 hours. A single dose would eliminate the need for a prescription for a drug like prednisone to hopefully improve compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55yo
* History of asthma
* Requires > 1 albuterol nebulizer
* Valid phone number

Exclusion Criteria:

* declines participation
* Past allergic reaction to corticosteroids
* Use of Oral steroids in the last 2 weeks
* Pregnant
* History of COPD, pulmonary fibrosis, cystic fibrosis, or other chronic lung disease
* History of HIV
* History of CHF
* History of Diabetes mellitus
* Active chickenpox (varicella) or shingles (herpes zoster)
* Active TB
* Requires admission to the Hospital
* Requires immediate airway intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2011-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Relapse for worsening asthma within 14 days of ED visit | 14-17 days
  Relapse will be defined as un unscheduled visit to see a doctor for worsening asthma within 14 days following their ED visit for asthma

SECONDARY OUTCOMES:
Compliance | 14 days
  Completion of study medications
Side effects | 14 days
  Assess if any side effects from the study medications
Symptoms persistence or improvement | 14-21 days
  Assessment of current rescue inhaler use and symptoms such as wheezing, cough, shortness of breath, and difficulty with activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Barry Simon, MD, Principal Investigator — Alameda County Medica Center
Locations (1):
- Alameda County Medical Center, Oakland, California, United States

REFERENCES:
- [Derived] Rehrer MW, Liu B, Rodriguez M, Lam J, Alter HJ. A Randomized Controlled Noninferiority Trial of Single Dose of Oral Dexamethasone Versus 5 Days of Oral Prednisone in Acute Adult Asthma. Ann Emerg Med. 2016 Nov;68(5):608-613. doi: 10.1016/j.annemergmed.2016.03.017. Epub 2016 Apr 22. PMID 27117874